CLINICAL TRIAL: NCT07240714
Title: Effects of a Web-based Support Programme for Cardiac Arrest Survivors: A Randomized Controlled Trial With Process Evaluation (The CARDIS Study)
Brief Title: Effects of an Web-based Support Programme for Cardiac Arrest Survivors
Acronym: CARDIS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Ingela Thylén, Assoc professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-06113-01
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Arrest (CA)
Keywords: Cardiac arrest; Digital support programme; Web-based intervention; Mental wellbeing; Quality of life; Fatigue; Cognitive function; Anxiety and depression; Post-traumatic stress; Randomized controlled trial; co-creation
MeSH Terms: conditions — Heart Arrest; Fatigue; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based Support Programme for Cardiac Arrest Survivors (Experimental)
  Interventions: Behavioral: Digital Support Programme
- Waitlist Control (Standard Care + Delayed Access) (No Intervention): Participants in this arm receive standard follow-up care according to national guidelines. They do not have access to the digital support programme during the study period. However, they are placed on a waitlist and are offered access to the programme after study completion.

INTERVENTIONS:
Behavioral: Digital Support Programme — The intervention consists of a web-based support programme designed for individuals recovering from cardiac arrest. Participants in the intervention group receive access to the programme for 12 weeks. The programme includes educational modules, patient and family stories, videos, practical exercises (e.g., breathing techniques, fatigue management), tools for personal recovery planning, and a moderated chat forum for peer support. Participants can access the content at their own pace and according to their individual needs. The programme is delivered entirely online and does not require any physical visits or clinical procedures.
  Arms: Web-Based Support Programme for Cardiac Arrest Survivors

SUMMARY:
The overall goal of this clinical trial is to learn if a web-based support programme can improve wellbeing in cardiac arrest survivors by helping them manage emotional, cognitive, and physical challenges. The study also explores how the programme is used and experienced in practice.

The main questions it aims to answer are:

* Can access to a web-based support programme improve overall wellbeing in cardiac arrest survivors?
* Can it also enhance quality of life, cognitive function, life satisfaction, and sleep, while reducing anxiety, depression, post-traumatic stress, and fatigue? Researchers will compare cardiac arrest survivors who receive a web-based support programme in addition to standard care with those who receive standard care alone, to see if the programme improves wellbeing and other health outcomes. After the study, the control group will also gain access to the programme.

Participants will:

* Be asked to complete online questionnaires at three time points: at the start of the study, after 3 months, and after 6 months.
* Be encouraged to use a web-based support programme for 3 months, with unlimited access, at their own pace and according to their individual needs (intervention group only).

DETAILED DESCRIPTION:
Cardiac arrest is a serious public health issue, affecting around 13,000 people annually in Sweden. Survivors often face long-term physical, cognitive, and emotional challenges, including anxiety, depression, fatigue, sleep disturbances, and post-traumatic stress. These difficulties can significantly impact daily life, and many survivors struggle to return to work or previous routines.

Although guidelines recommend follow-up within 1-3 months after hospital discharge, support is often fragmented and varies across regions. Survivors frequently report limited access to reliable information and emotional support. Research has shown that structured education and rehabilitation are essential for both survivors and their families, yet current care models rarely address these needs in a comprehensive way.

To help fill this gap, a web-based support programme was co-created in 2024-2025 by researchers, healthcare professionals, cardiac arrest survivors, and patient organizations. The programme includes educational modules, patient and family stories, videos, practical exercises, and tools for self-management and personal recovery planning. It also features a moderated chat forum for peer support. A feasibility study showed that the programme was easy to use and perceived as relevant and helpful.

The study begins with a pilot phase (n=10) to test study procedures, followed by a randomized controlled trial (RCT) with 120 participants across eight Swedish regions. Participants are recruited during routine follow-up visit one month after discharge. All participants receive standard care. Those randomized to the intervention group gain access to the digital support programme for 12 weeks. The control group receives standard care and gains access to the programme after study completion.

Consent and data collection are handled digitally. Participants are asked to complete online surveys at baseline, 3 months, and 6 months. These surveys cover wellbeing, quality of life, sleep, fatigue, emotional health, and cognitive function. The study also collects usage data from the programme to understand how participants engage with the content. No physical tests or extra clinic visits are required.

The study aims to generate new knowledge about how digital tools can support recovery after cardiac arrest, improve wellbeing, and reduce healthcare burden by offering accessible, person-centered rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Survival of a cardiac arrest 1 to 3 months prior to enrollment
* Access to a mobile phone, tablet, or computer with internet connection

Exclusion Criteria:

* Insufficient language or cognitive ability to engage with a digital intervention and complete questionnaires in Swedish
* Participation in another study involving the collection of patient-reported outcome measures (PROMs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Overall Wellbeing at 3 months. | From baseline to 3 months after enrollment.
  The Questionnaire on Well-Being is a tool designed to capture subjective well-being. It consists of 18 questions, each rated from 0 to 4, which are added together to give a total score between 0 and 72. Higher scores reflect greater perceived well-being, while scores below 50 have been linked to significant psychological distress.

SECONDARY OUTCOMES:
Change from Baseline in Quality of Life at 3 and 6 months. | From baseline to 3 and 6 months after enrollment.
  Change from baseline in Quality of Life (EuroQol Five-Dimension Five-Level questionnaire, EQ-5D-5L).
  Score range: 0 to 1 (index value). Higher scores indicate better quality of life.
  Change from baseline in Quality of Life (EuroQol Visual Analogue Scale). Score range: 0 to 100. Higher scores indicate better self-rated health.
  Outcomes will be analyzed both as change from baseline to each time point (3 and 6 months), and as within-subject change between the 3- and 6-months assessments to evaluate sustained or delayed effects of the intervention.
Change from baseline in Life Satisfaction at 3 and 6 months. | From baseline to 3 and 6 months after enrollment.
  Change from baseline in Life Satisfaction (Life Satisfaction Questionnaire, LiSat-11) at 3 and 6 months.
  Score range: 11 to 66. Higher scores indicate greater life satisfaction. Outcomes will be analyzed both as change from baseline to each time point (3 and 6 months), and as within-subject change between the 3- and 6-months assessments to evaluate sustained or delayed effects of the intervention.
Change from baseline in Anxiety at 3 and 6 months. | From baseline to 3 and 6 months after enrollment.
  Change from baseline in Anxiety (Generalised Anxiety Disorder 7-item scale, GAD-7) at 3 and 6 months.
  Score range: 0 to 21. Higher scores indicate more severe anxiety symptoms.
  Outcomes will be analyzed both as change from baseline to each time point (3 and 6 months), and as within-subject change between the 3- and 6-months assessments to evaluate sustained or delayed effects of the intervention.
Change from baseline in Depression at 3 and 6 months. | From baseline to 3 and 6 months after enrollment.
  Change from baseline in Depression (Patient Health Questionnaire 9-item scale, PHQ-9) at 3 and 6 months. Score range: 0 to 27. Higher scores indicate more severe depressive symptoms.
  Outcomes will be analyzed both as change from baseline to each time point (3 and 6 months), and as within-subject change between the 3- and 6-months assessments to evaluate sustained or delayed effects of the intervention.
Change from baseline in Post-Traumatic Stress at 3 and 6 months. | From baseline to 3 and 6 months after enrollment.
  Change from baseline in Post-Traumatic Stress (Impact of Event Scale - Revised, IES-R) at 3 and 6 months. Score range: 0 to 88. Higher scores indicate more severe post-traumatic stress symptoms.
  Outcomes will be analyzed both as change from baseline to each time point (3 and 6 months), and as within-subject change between the 3- and 6-months assessments to evaluate sustained or delayed effects of the intervention.
Change from baseline in Fatigue at 3 and 6 months. | From baseline to 3 and 6 months after enrollment.
  Change from baseline in Fatigue (Modified Fatigue Impact Scale, MFIS-21) at 3 and 6 months. Score range: 0 to 84. Higher scores indicate greater impact of fatigue.
  Outcomes will be analyzed both as change from baseline to each time point (3 and 6 months), and as within-subject change between the 3- and 6-months assessments to evaluate sustained or delayed effects of the intervention.
Change from baseline in Sleep at 3 and 6 months. | From baseline to 3 and 6 months after enrollment.
  Change from baseline in Sleep (Minimal Insomnia Symptom Scale, MISS) at 3 and 6 months. Score range: 0 to 12. Higher scores indicate more severe insomnia symptoms.
  Outcomes will be analyzed both as change from baseline to each time point (3 and 6 months), and as within-subject change between the 3- and 6-months assessments to evaluate sustained or delayed effects of the intervention.
Change from baseline in Cognitive Function at 3 and 6 months. | From baseline to 3 months after enrollment.
  Change from baseline in Cognitive Function (single-item question on perceived cognitive difficulties) at 3 and 6 months. Score range: 1 to 5. Higher scores indicate greater perceived cognitive impairment.
  Outcomes will be analyzed both as change from baseline to each time point (3 and 6 months), and as within-subject change between the 3- and 6-months assessments to evaluate sustained or delayed effects of the intervention.

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Dept of Cardiology, Linköping
  - Dept of Cardiology, Motala
  - Dept of Cardiology, Norrköping

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available to members of the research team after the principal investigator has completed blinded analyses of the primary and secondary outcomes. Data will be stored securely and access will be restricted to authorized collaborators under data use agreements.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning after completion of the blinded primary and secondary outcome analyses by the principal investigator, with no defined end date.
Access Criteria: Access to de-identified individual participant data (IPD) will be granted to members of the research team after completion of the blinded analysis of primary and secondary outcomes by the principal investigator. Each researcher must submit a brief description of the planned analyses and sign a data use agreement outlining responsibilities for data handling, confidentiality, and publication ethics. Access requests will be reviewed and approved by the principal investigator.